CLINICAL TRIAL: NCT02949856
Title: Endotracheal Tube Intracuff Pressure Change After Changing Position From Neutral to Hyperextension of Neck - Comparison of a Tapered Shaped- and Cylindrical Shaped Cuff
Brief Title: E-T Tube Cuff Pressure Change After Changing Position From Neutral to Hyperextension of Neck
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-05-032-001
Record Dates: First submitted 2016-10-20; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Thyroidectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tapered (Experimental): Mallinckrodt, COVIDIEN
  Interventions: Device: Mallinckrodt, COVIDIEN
- Cylindrical (Active Comparator): Endotracheal tube, Unomedical
  Interventions: Device: Endotracheal tube, Unomedica

INTERVENTIONS:
Device: Mallinckrodt, COVIDIEN
  Arms: Tapered
Device: Endotracheal tube, Unomedica
  Arms: Cylindrical

SUMMARY:
This study evaluates difference of the endotracheal tube cuff pressure between a tapered- versus a cylindrical- shaped cuff after changing from neutral to hyperextension of neck.

Fifty patients undergoing thyroidectomy are randomly allocated into two groups (tapered- and cylindrical-shaped cuff). Endotracheal tube cuff pressure is initially set at 20 cmH20 in the supine neutral position and is measured after the change to the neck extension.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical classification 1-3, 18-70 year old, thyroidectomy

Exclusion Criteria:

* difficult intubation, history of cervical disease, motion limitation of neck, morbid obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in intracuff pressure | 1 year

SECONDARY OUTCOMES:
Change in distance from carina to tip of tube | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Cheol Lee, MD, PhD, Principal Investigator — Keimyung University Dongsan Medical Center

IPD SHARING:
Plan to Share IPD: No